CLINICAL TRIAL: NCT06989242
Title: Yoga-based, Movement Therapy Device as Noninvasive Glymphatic Clearance Augmentation in Alzheimer's Disease. The Feasibility and Safety Trial With Preliminary Clinical, Digital, and Fluid Biomarker Proxies of Glymphatic Clearance
Brief Title: Yoga-based, Movement Therapy Device as Noninvasive Glymphatic Clearance Augmentation in Alzheimer's Disease.
Acronym: ReGlyde
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CIATRIX, INC. (Industry)
Collaborators: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG-CZSK-PH2; RG-CZSK-PH2 (Other: CIATRIX Inc.)
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment (MCI)
Keywords: Mind-Body Intervention; Medical Device; CSF flow; fNIRS; Feasibility Study; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single-arm interventional feasibility and safety study evaluating a yoga-based therapeutic device in individuals diagnosed with Alzheimer's disease (stages 3 and 4). The intervention combines guided movement and rhythmic breathing. The study assesses feasibility, safety, and preliminary effects on cognitive function, physiological markers (e.g., fNIRS, HRV, posture), and fluid biomarkers.
Masking Description: No other parties who are masked are involved in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention Arm - Device-Guided Movement and Breathing (Experimental): Participants in this arm will receive a yoga-based intervention delivered through a powered therapeutic device that guides rhythmic breathing and spinal movement. The intervention is designed to mimic traditional yoga poses such as Marjariasana (cat-cow) and is conducted over multiple sessions. The study aims to assess feasibility, safety, and preliminary effects on cognitive function, physiological measures (e.g., fNIRS, HRV, posture), and fluid biomarkers in individuals with Alzheimer's disease (stages 3 and 4).
  Interventions: Device: Yoga-Based Therapeutic Device (incorporating guided breathing and movement)

INTERVENTIONS:
Device: Yoga-Based Therapeutic Device (incorporating guided breathing and movement) — The Fluere™ Therapeutic Device is a computer-guided, electro-mechanical system designed to simulate yoga-inspired spinal movement and rhythmic breathing. Resembling a dental chair, the device dynamically adjusts spinal curvature to replicate motion patterns associated with deep abdominal breathing, similar to Kundalini or Qi Gong breathwork. The device operates automatically, with optional manual adjustments by the researcher.
  Other Names: Rhythmic Breathing and Spinal Mobilization Chair

SUMMARY:
This clinical trial evaluates a yoga-based intervention delivered through a powered therapeutic device designed to guide breathing and body movements. Building on evidence that mind-body practices may promote healthy aging, cognitive function, and glymphatic flow, the study uses physiological measurements, including fNIRS and wearable sensors, to investigate mechanisms and potential benefits in individuals at risk for Alzheimer's disease.

DETAILED DESCRIPTION:
Brief Summary:

The current trial builds on recent findings that highlight the effectiveness of mind-body interventions, such as yoga and deep abdominal breathing, in promoting healthy aging and slowing cognitive decline. Research suggests that yoga and body-mind practices can improve well-being and reduce biological markers of aging in both healthy older adults and those at risk for dementia. Yogic breathing and body movements may enhance cerebrospinal fluid (CSF) flow as an important component of the glymphatic function. The trial employs physiological measurements, including fNIRS and wearable sensors, to investigate the mechanisms and clinical benefits of yoga-based interventions for AD.

The primary objective is to assess the safety, tolerability, feasibility of a 4-week Fluere™ therapy protocol for stage 3 and 4 AD patients.

The secondary objectives focus on clinical effectiveness related to:

1. Body posture improvement
2. Changes in HRV (reflecting the stress level and quality of sleep)

Although the duration of the study is short, and the study is not powered to detect changes in biomarkers or clinical efficacy, secondary endpoints will be analyzed to assess trends in improvement from baseline.

Additional secondary outcomes will focus on biomarker proxies of glymphatic clearance:

1. Impact on digital biomarkers (neuro-fluid dynamics (hemodynamics, CSF) and redox state of cytochrome-c-oxidase activity using fNIRS)
2. Effect on plasma biomarkers associated with neurodegeneration, inflammation and neural plasticity - GFAP, NfL and S100B and BDNF
3. Cognitive (spatial memory) and functional outcomes
4. Sleep patterns and quality through wearable devices and questionnaires

ELIGIBILITY:
Inclusion Criteria:

* 55-85 years of age
* Current diagnostic criteria for stage 3 AD patients (AD-MCI)
* Current diagnostic criteria for stage 4 AD patients (mAD)
* Able to provide consent to be in the study
* Willing and able to participate in study activities
* Able to lay supine for 30-45 minutes
* Able to walk 20 meters
* Willing to not perform additional mind-body practices during the duration of the study
* Able to use a wearable electronic device (Smart watch)

Exclusion Criteria:

* Inability to provide informed consent
* Regular use of muscle relaxants or anti-anxiety drugs
* Any muscle or skeletal issues that would make it difficult to lie still in the supine position for the 1-hour physical therapy
* Craniospinal disorders, e.g., Chiari Malformation.
* Spinal injuries, clinically relevant disc herniation, spinal stenosis, spondylolisthesis in the sacral, lumbar, thoracic, or cervical spine, spinal bifida, Recent Spinal Surgery
* Severe osteoporosis with a risk of fracture
* History of neurological disorders such as stroke (during the last year before study start), mild brain injury within past 6 months, multiple sclerosis, presence of intracranial hemorrhage, hydrocephalus, meningitis, encephalitis, brain tumor (except of asymptomatic meningioma GI)
* Serious sleep disorders - narcolepsy
* Major or uncontrolled psychiatric illness or major depression.
* Any condition requiring the use of medication that acts on the brain such as stimulants, sedatives (hypnotics and benzodiazepines), antipsychotics, and anti-anxiety medications, (we will include patients with stable antidepressant treatment and being on mild anti-seizure medication due to polyneuropathy)
* Active infection or uncontrolled significant systemic illnesses
* Asthma, chronic obstructive pulmonary disease
* Recent hearth attack, Implantable defibrillator, poorly controlled blood pressure cardiac arrhythmia, unstable angina pectoris, or symptomatic congestive heart failure
* People at risk of blood clots or deep vein thrombosis (DVT) might want to avoid prolonged sitting in the chair
* Obesity over 135 kg (300lb)
* Smoking more than 5 cigarettes a day or drinking more than 1 alcoholic beverage a day

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number and type of intervention-related adverse events as assessed by a yoga-specific adverse events questionnaire | Throughout the 4-week intervention period
  Safety will be evaluated using a standardized yoga-specific adverse events questionnaire administered after each session. Adverse events will be recorded, categorized (e.g., musculoskeletal, autonomic, psychological), and summarized by frequency and severity. Only events judged as related to the intervention will be included.
Number of participants completing ≥90% of scheduled intervention sessions | 4 weeks (intervention period)
  Feasibility of the intervention will be assessed by the number of participants who attend at least 90% of scheduled sessions (i.e., ≥11 out of 12 sessions). Reported as count and percentage of total enrolled participants.
Mean percentage of completed intervention sessions per participant | 4 weeks (intervention period)
  Calculated as the average percentage of completed sessions per participant across the study population. This reflects session adherence at the group level.
Number of participants who withdraw from the study before completing intervention | 4 weeks (intervention period)
  The dropout rate will be determined by the number of participants who discontinue the study before completing all planned sessions, regardless of reason.

SECONDARY OUTCOMES:
Change in Heart Rate Variability During Therapy over time | During each session across 4 weeks
  HRV is measured during device-guided breathing and movement sessions using wearable sensors.
Change in vertical postural alignment as measured by digital posture analysis | Baseline and 4 timepoints altogether corresponding to 4 treatment weeks
  Posture will be quantified using photographic images captured weekly, with a standardized posture grid overlaid on each image. The grid will allow for objective measurement of spinal alignment and the sagittal vertical axis.
Change in spine flexibility as measured by the Thomayer test (in cm) | Baseline and weekly
  Spine flexibility will be assessed using the Thomayer forward bend test. Participants reach toward the floor from a standing position with knees straight, and the distance between fingertips and floor (positive or negative) will be recorded and compared pre/post.
Change in nightly average heart rate variability (SMSSD) during sleep as measured by wearable sensors in Milliseconds (ms) | Nightly, throughout the 4-week study period
  HRV will be continuously monitored using validated wearable PPG-based devices. The nightly average root mean square of successive differences (RMSSD) will be extracted and averaged weekly. Baseline-week values will be compared to Week 4 values.
Change in nightly average resting heart rate during sleep as measured by wearable sensors (in bpm) | Nightly, throughout the 4-week study period
  Resting heart rate will be measured each night using wearable devices during sleep. Weekly averages will be calculated and compared from baseline to Week 4.
Change in nightly average respiratory rate (Breaths per minute) during sleep as measured by wearable sensors | Nightly, throughout the 4-week study period
  Respiratory rate will be assessed via wearable sensors each night during sleep. Weekly averages will be calculated and compared between baseline and the end of the intervention.
Change in cortical hemodynamic activity (HbO and HbR concentrations) at rest and during intervention, measured by fNIRS | Baseline, Week 4, and during each intervention session
  Hemodynamic changes will be assessed using fNIRS to measure oxygenated (HbO) and deoxygenated hemoglobin (HbR) concentrations in the prefrontal cortex.
Change in cortical water signal (tissue hydrodynamics) measured by H2O-specific wavelength sensor | Baseline, Week 4, and during each intervention session
  Hydrodynamic properties of cortical tissue will be assessed using NIR absorption at water-sensitive wavelengths (e.g., ~980 nm). Water content changes will be used as a proxy for CSF bulk flow / interstitial flow.
Change in oxidation state of cytochrome c oxidase measured by broadband fNIRS | Baseline, Week 4, and during each intervention session
  Redox activity of mitochondrial cytochrome c oxidase (oxCCO) will be evaluated using broadband fNIRS to assess metabolic shifts in the prefrontal cortex.
Change in nightly sleep stage distribution as measured by PPG-based wearable sensors - Percentage of total sleep time in each of the sleep stages | Nightly, over the 4-week intervention period
  Sleep architecture will be measured using photoplethysmography-based wearable devices each night. Proportions of time spent in light, deep, and REM sleep will be computed and averaged weekly.
Change in sleep quality subscale score (B-PSQI) from the GlymphActive Questionnaire | Baseline and Week 4
  Sleep quality will be assessed using the B-PSQI subscale of the GlymphActive Questionnaire, which includes the 7 standard components of the PSQI-B. Total scores range from 0 to 21, with higher scores indicating worse sleep quality. Score (range 0-21; higher = worse sleep quality)
Change in spatial navigation performance (corrent responses) as measured by the Intersections Spatial Memory Cognitive Task | Familiarization at screening, Baseline and Week 4
  The Intersections Task is a 3D computerized spatial navigation test mimicking real-city routes. It assesses egocentric and allocentric spatial memory and perspective-taking. Participants are transported across intersections during the learning phase and later asked to recall correct routes.
Change in global cognitive function as measured by the Mini-Mental State Examination (MMSE) | Baseline and at Week 4
  Global cognitive function will be assessed using the MMSE. This brief screening tool evaluates orientation, memory, attention, language, and visuospatial skills. Scores range from 0 to 30. Higher scores indicate better cognitive function. Score (range 0-30; higher = better cognition)
Change in functional ability as measured by the Functional Activities Questionnaire (FAQ-CZ) | Baseline and at Week 4
  Functional status will be assessed using the Czech version of the FAQ-CZ, which evaluates the participant's ability to perform instrumental activities of daily living. Higher scores indicate greater functional impairment. Score (range 0-30; higher = more impairment)
Change in subjective memory complaints as measured by the McNair Memory Complaint Questionnaire | Baseline and Week 4
  Subjective memory will be evaluated using the McNair Memory Complaint Questionnaire. It assesses the frequency and severity of self-perceived memory problems in daily life. Higher scores reflect more frequent complaints. The questionnaire consists of 21 items assessing the frequency and severity of perceived memory problems in everyday life. Each item is rated on a 5-point Likert scale. Total scores range from 0 to 84, with higher scores indicating more frequent or severe memory complaints. Score (range 0-84; higher = worse subjective memory)
Change in anxiety symptoms as measured by the Beck Anxiety Inventory (BAI) | Baseline and Week 4
  Anxiety symptoms will be assessed using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire designed to measure the severity of anxiety in adults. Each item is scored on a 0-3 scale, resulting in a total score range from 0 to 63. Higher scores indicate greater anxiety severity. Score (range 0-63; higher = worse anxiety)
Change in depressive symptoms as measured by the Geriatric Depression Scale - Short Form (GDS-15) | Baseline and Week 4
  Depressive symptoms will be assessed using the 15-item version of the Geriatric Depression Scale (GDS-15). This self-report tool consists of yes/no questions focused on mood, motivation, and daily functioning. Total scores range from 0 to 15, with higher scores indicating greater depressive symptom severity. Score (range 0-15; higher = worse depression)
Change in Global QoL score as measured by the WHOQOL-BREF | Baseline and Week 4
  Global quality of life and general health will be assessed using the first two items of the WHOQOL-BREF questionnaire. Participants rate their overall quality of life and satisfaction with health. Scores are averaged and transformed to a 0-100 scale. Higher scores indicate better perceived overall well-being and health.
Change in plasma neurofilament light chain (NfL) concentration | Baseline and Week 4
  Neurofilament light chain, a biomarker of axonal damage, will be measured in plasma using ultra-sensitive SIMOA technology. Concentrations at baseline and Week 4 will be compared to assess neurodegeneration-related changes. Unit of measure: Picograms per milliliter (pg/mL)
Change in plasma brain-derived neurotrophic factor (BDNF) concentration | Baseline and Week 4
  Plasma levels of BDNF will be quantified using SIMOA technology. BDNF is a neurotrophin involved in neuroplasticity and synaptic maintenance. Pre-/post-intervention levels will be compared. Unit of Measure: Nanograms per milliliter (ng/mL)
Change in plasma glial fibrillary acidic protein (GFAP) concentration | Baseline and Week 4
  GFAP, a marker of astrocytic activity and gliosis, will be measured in plasma using SIMOA. Baseline and Week 4 concentrations will be compared to assess glial response to intervention. Picograms per milliliter (pg/mL) as units of measure.
Change in plasma S100 calcium-binding protein B (S100B) concentration | Baseline and Week 4
  S100B, a glial-derived protein associated with neuroinflammation and blood-brain barrier dysfunction, will be measured using SIMOA. Changes between baseline and Week 4 will be analyzed. Nanograms per milliliter (ng/mL) as units of measure

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Simko, MA. PhD., Study Director — Masaryk University, The International Clinical Research Center of St. Anne's University Hospital in Brno (FNUSA-ICRC), CIATRIX Inc.; Katerina Sheardova, MD. PhD., Principal Investigator — The International Clinical Research Center of St. Anne's University Hospital in Brno (FNUSA-ICRC)
Locations (3):
- Czechia (2):
  - Neuro Health Centrum S.R.O, Brno
  - Neuropsychiatrie s.r.o., Terronska 580/19, Prague
- AuraMedica s.r.o., Neurologická ambulancia, OMNIA BUSINESS CENTER, Tomášikova 19081/28C, Bratislava, Slovakia, Slovakia

REFERENCES:
- See also: Related Info — https://www.ciatrix.com/